CLINICAL TRIAL: NCT03981835
Title: Management of Antiplatelet Regimen During Surgical Procedures (MARS Registry)
Brief Title: Management of Antiplatelet Regimen During Surgical Procedures
Acronym: MARS
Status: Completed | Type: Observational
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: STU-2018-0398
Record Dates: First submitted 2019-06-06; First posted 2019-06-11 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2023-12

CONDITIONS: Cardiac Surgery; Surgery; Percutaneous Coronary Intervention; Surgery--Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Post -PCI Patients scheduled for Cardiac Surgery: Post -PCI Patients (PCI within the last 2 years) who are currently on Dual- Antiplatelet (DAPT) Medication or have a current indication for DAPT, who will be undergoing Cardiac Surgery. No intervention will be administered.
- Post -PCI Patients scheduled for Non- Cardiac Surgery: Post -PCI Patients (PCI within the last 2 years) who are currently on Dual- Antiplatelet (DAPT) Medication or have a current indication for DAPT, who will be undergoing Non-Cardiac Surgery. No intervention will be administered.

SUMMARY:
There are key differences today in clinical practice regarding perioperative management of post-PCI patients on DAPT undergoing NCS. Moreover, there are significant differences between bridging agents, and improved safety of current-generation DES. Given the significant limitations of current studies a well-designed registry to study current U.S. practice patterns and the bleeding or ischemic risks associated with the various perioperative DAPT management strategies including bridging and no bridging will significantly add to the understanding of the current problem and associated risks of patients. These data could form the basis for conducting future randomized clinical trials (RCTs) in this area. NCS in post-PCI patients on chronic DAPT presents a complex interaction of both ischemic and bleeding risks.

The MARS registry will study the area of perioperative antiplatelet therapy management through a multicenter observational national registry designed to collect pre-operative, intra-operative and post-operative clinical strategies, therapeutic interventions and outcomes data. This proposal outlines the role of a highly experienced clinical trial team to conduct a multicenter prospective registry. This question is highly relevant to a diverse group of medical providers and millions of patients in the US and around the world; this will be the first such U.S. registry to address this critically important public health issue.

Study objectives:

i. To collect data on contemporary clinical practice in the U.S. on managing post percutaneous coronary intervention (PCI) DAPT in patients scheduled to undergo NCS and CS.

ii. To assess ischemic and bleeding endpoints in this group of patients during the study period.

iii. To generate initial data to plan for future large-scale randomized clinical trials on perioperative management of DAPT.

DETAILED DESCRIPTION:
1. Registry infrastructure: The proposed registry is a multicenter prospective registry that is designed to capture perioperative DAPT management strategies in patients undergoing NCS or CS post-PCI. It will be adjudicated and monitored for data accuracy and completeness. The registry will be de-identified and compliant with HIPPA regulations and will be located on secure servers of the University of Texas Southwestern Medical Center (UTSW). Full-time staff that includes an information technology officer and data programmer manages the registry servers professionally. The servers are backed up daily and provide on-line secure access to site investigators and coordinators. The current registry structure is already in use for a national peripheral artery disease registry and can be viewed at www.XLPAD.org. The MARS registry will include two separate registry arms to capture data on two distinct cohorts: (i) NCS and (ii) CS.
2. Hypothesis: This observational registry is designed to test whether 30-day NACE associated with IV APT bridging is ≥6%.
3. Study period: period of 14 days prior to surgery to 30 days post-surgery.
4. Study eligible NCS or CS :

   * Study eligible non-cardiac surgeries and procedures:

     1. Intra-abdominal surgery (e.g., bowel or visceral organ resection) *
     2. Intra-thoracic surgery (e.g., lung resection) *
     3. Major orthopedic surgery (e.g., hip or knee replacement)
     4. Peripheral arterial revascularization (e.g., aortic aneurysm repair*, vascular bypass*, carotid surgery)
     5. Urologic surgery (e.g., prostatectomy*, bladder tumor resection);
     6. Major procedure (e.g., renal, lung or liver transplants*, biopsy of lung, head and neck surgery*)
     7. Breast and other surgeries or procedures requiring DAPT interruption as per the clinical team *High-risk NCS, remaining classified as low-intermediate
   * Study eligible cardiac surgeries and procedures

     1. Coronary artery bypass graft (CABG)
     2. Cardiac valve repair or replacement with or without CABG
     3. Surgical arrhythmia treatment (MAZE procedure)
     4. Pericardial procedures
     5. Thoracoscopic procedures
     6. Other cardiothoracic procedures (please contact study tem)
5. Study population: Post-PCI patients on DAPT undergoing NCS and CS. Patients will be asked to sign an informed consent form (ICF) or ICF deferred based on the mandate of their respective institutional review boards (IRB).
6. Registry data collection: The registry will be built on the NHLBI's REDCap data collection portal that is available to UTSW under an Academic Information Systems NIH grant UL1-RR024982. The proposed MARS Registry data collection portal. The data collection portal has been designed to facilitate comprehensive data collection from 2 weeks prior to surgery to 30±7 days post-surgery and includes demographics, laboratory, coronary revascularization, medication and clinical outcome information. Baseline information will include demographic, relevant medical history, preoperative medications and laboratory values and any preoperative clinical events during the study period. Procedure related data will include surgical procedure details, intraoperative medications and medications, laboratory values and clinical outcomes from the day of surgery till hospital discharge. Postoperative data collection will include medications, laboratory values and clinical events between hospital discharge and 30 days post-discharge. Data will be entered into a secure and HIPPA compliant online REDCap data collection portal. No study related procedures, interventions or follow-ups are required. Each site staff will enter data based on electronic health records (EHR), which wills serve as the primary data source. Out of hospital medical records will need to be incorporated or documented as part of a given participants' source data. All participants will be given the opportunity to re-evaluate their decisions regarding participation in the MARS Registry. The MARS registry will include two separate arms of the registry to capture data on two distinct cohorts: (i) NCS and (ii) CS.

ELIGIBILITY:
Inclusion Criteria:

* Patients with PCI within the past 2 years who: a. Are currently on DAPT, OR b. Have a current indication for DAPT
* Scheduled for NCS or CS.
* Willing and able to provide an informed consent (if needed based on institutional IRB requirements).

Exclusion Criteria:

* Emergent (6 hours) surgery post-PCI on DAPT that precludes a thorough informed consent process.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Post-PCI patients on DAPT undergoing NCS and CS. Patients will be asked to sign an informed consent form (ICF) based on the mandate of their respective institutional review boards (IRB).
Sampling Method: Non-Probability Sample
Enrollment: 147 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Rate of Net adverse cardiovascular events (NACE) over the study period | 2 weeks prior to surgery to up to 30 days post-surgery
  A composite of cardiovascular (CV) death, non-fatal myocardial infarction (MI), ischemic stroke, need for urgent coronary revascularization (UCR) or Bleeding Academic Research Consortium (BARC) ≥3 bleeding during the study period.

SECONDARY OUTCOMES:
Incidence of individual components of NACE over the study period | 2 weeks prior to surgery to up to 30 days post-surgery
  Incidence of cardiovascular (CV) death, non-fatal myocardial infarction (MI), ischemic stroke, need for urgent coronary revascularization (UCR) or Bleeding Academic Research Consortium (BARC) ≥3 bleeding during the study period.
Incidence of IV antiplatelet (APT) bridging and comparison of IV APT bridging and no bridging strategies. | 2 weeks prior to surgery to up to 30 days post-surgery
  Incidence of IV antiplatelet (APT) bridging and comparison of IV APT bridging and no bridging strategies.
Time to NACE | 2 weeks prior to surgery to up to 30 days post-surgery
  Time to NACE
All-cause mortality | 2 weeks prior to surgery to up to 30 days post-surgery
  All-cause mortality
Incidence of definite and probable stent thrombosis (ST). | 2 weeks prior to surgery to up to 30 days post-surgery
  Incidence of definite and probable stent thrombosis (ST).
Length of hospital stay (LOS). | 2 weeks prior to surgery to up to 30 days post-surgery
  Length of hospital stay (LOS).
Health economic analysis comparing cost-effectiveness of IV APT bridging and no bridging strategies. | 2 weeks prior to surgery to up to 30 days post-surgery
  Health economic analysis comparing cost-effectiveness of IV APT bridging and no bridging strategies.

CONTACTS AND LOCATIONS:
Overall Officials: Subhash Banerjee, MD, Study Chair — Baylor Scott & White Research Institute
Locations (5):
- United States (5):
  - University of Florida, Jacksonville, Florida
  - Dallas VA Medical Center, Dallas, Texas
  - Baylor Scott & White Research Institute, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Mary Washington Hospital, Fredericksburg, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Auerbach DI, Maeda JL, Steiner C. Hospital Stays with Cardiac Stents, 2009. 2012 Apr. In: Healthcare Cost and Utilization Project (HCUP) Statistical Briefs [Internet]. Rockville (MD): Agency for Healthcare Research and Quality (US); 2006 Feb-. Statistical Brief #128. Available from http://www.ncbi.nlm.nih.gov/books/NBK97358/ PMID 22696778
- [Background] Bangalore S, Gupta N, Guo Y, Feit F. Trend in the use of drug eluting stents in the United States: insight from over 8.1 million coronary interventions. Int J Cardiol. 2014 Jul 15;175(1):108-19. doi: 10.1016/j.ijcard.2014.04.269. Epub 2014 May 9. PMID 24852837
- [Background] Levine GN, Bates ER, Blankenship JC, Bailey SR, Bittl JA, Cercek B, Chambers CE, Ellis SG, Guyton RA, Hollenberg SM, Khot UN, Lange RA, Mauri L, Mehran R, Moussa ID, Mukherjee D, Nallamothu BK, Ting HH; ACCF; AHA; SCAI. 2011 ACCF/AHA/SCAI Guideline for Percutaneous Coronary Intervention: executive summary: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines and the Society for Cardiovascular Angiography and Interventions. Catheter Cardiovasc Interv. 2012 Feb 15;79(3):453-95. doi: 10.1002/ccd.23438. No abstract available. PMID 22328235
- [Background] Capodanno D, Angiolillo DJ. Management of antiplatelet therapy in patients with coronary artery disease requiring cardiac and noncardiac surgery. Circulation. 2013 Dec 24;128(25):2785-98. doi: 10.1161/CIRCULATIONAHA.113.003675. No abstract available. PMID 24366588
- [Background] Bonaca MP, Braunwald E, Sabatine MS. Long-Term Use of Ticagrelor in Patients with Prior Myocardial Infarction. N Engl J Med. 2015 Sep 24;373(13):1274-5. doi: 10.1056/NEJMc1508692. No abstract available. PMID 26398078
- [Background] Alshawabkeh LI, Prasad A, Lenkovsky F, Makary LF, Kandil ES, Weideman RA, Kelly KC, Rangan BV, Banerjee S, Brilakis ES. Outcomes of a preoperative "bridging" strategy with glycoprotein IIb/IIIa inhibitors to prevent perioperative stent thrombosis in patients with drug-eluting stents who undergo surgery necessitating interruption of thienopyridine administration. EuroIntervention. 2013 Jun 22;9(2):204-11. doi: 10.4244/EIJV9I2A35. PMID 23454910
- [Background] Habib A, Finn AV. Endothelialization of drug eluting stents and its impact on dual anti-platelet therapy duration. Pharmacol Res. 2015 Mar;93:22-7. doi: 10.1016/j.phrs.2014.12.003. Epub 2014 Dec 19. PMID 25533811
- [Background] McFadden EP, Stabile E, Regar E, Cheneau E, Ong AT, Kinnaird T, Suddath WO, Weissman NJ, Torguson R, Kent KM, Pichard AD, Satler LF, Waksman R, Serruys PW. Late thrombosis in drug-eluting coronary stents after discontinuation of antiplatelet therapy. Lancet. 2004 Oct 23-29;364(9444):1519-21. doi: 10.1016/S0140-6736(04)17275-9. PMID 15500897
- [Background] Ong AT, Hoye A, Aoki J, van Mieghem CA, Rodriguez Granillo GA, Sonnenschein K, Regar E, McFadden EP, Sianos G, van der Giessen WJ, de Jaegere PP, de Feyter P, van Domburg RT, Serruys PW. Thirty-day incidence and six-month clinical outcome of thrombotic stent occlusion after bare-metal, sirolimus, or paclitaxel stent implantation. J Am Coll Cardiol. 2005 Mar 15;45(6):947-53. doi: 10.1016/j.jacc.2004.09.079. PMID 15766834
- [Background] Regar E, Lemos PA, Saia F, Degertekin M, Tanabe K, Lee CH, Arampatzis CA, Hoye A, Sianos G, de Feyter P, van der Giessen WJ, Smits PC, van Domburg RT, Serruys PW. Incidence of thrombotic stent occlusion during the first three months after sirolimus-eluting stent implantation in 500 consecutive patients. Am J Cardiol. 2004 May 15;93(10):1271-5. doi: 10.1016/j.amjcard.2004.02.013. PMID 15135702
- [Background] Iakovou I, Schmidt T, Bonizzoni E, Ge L, Sangiorgi GM, Stankovic G, Airoldi F, Chieffo A, Montorfano M, Carlino M, Michev I, Corvaja N, Briguori C, Gerckens U, Grube E, Colombo A. Incidence, predictors, and outcome of thrombosis after successful implantation of drug-eluting stents. JAMA. 2005 May 4;293(17):2126-30. doi: 10.1001/jama.293.17.2126. PMID 15870416
- [Background] Rossini R, Musumeci G, Capodanno D, Lettieri C, Limbruno U, Tarantini G, Russo N, Calabria P, Romano M, Inashvili A, Sirbu V, Guagliumi G, Valsecchi O, Senni M, Gavazzi A, Angiolillo DJ. Perioperative management of oral antiplatelet therapy and clinical outcomes in coronary stent patients undergoing surgery. Results of a multicentre registry. Thromb Haemost. 2015 Feb;113(2):272-82. doi: 10.1160/TH14-05-0436. Epub 2014 Oct 2. PMID 25274620
- [Background] Silber S, Kirtane AJ, Belardi JA, Liu M, Brar S, Rothman M, Windecker S. Lack of association between dual antiplatelet therapy use and stent thrombosis between 1 and 12 months following resolute zotarolimus-eluting stent implantation. Eur Heart J. 2014 Aug 1;35(29):1949-56. doi: 10.1093/eurheartj/ehu026. Epub 2014 Feb 7. PMID 24510638
- [Background] Fleisher LA, Fleischmann KE, Auerbach AD, Barnason SA, Beckman JA, Bozkurt B, Davila-Roman VG, Gerhard-Herman MD, Holly TA, Kane GC, Marine JE, Nelson MT, Spencer CC, Thompson A, Ting HH, Uretsky BF, Wijeysundera DN. 2014 ACC/AHA guideline on perioperative cardiovascular evaluation and management of patients undergoing noncardiac surgery: executive summary: a report of the American College of Cardiology/American Heart Association Task Force on practice guidelines. Developed in collaboration with the American College of Surgeons, American Society of Anesthesiologists, American Society of Echocardiography, American Society of Nuclear Cardiology, Heart Rhythm Society, Society for Cardiovascular Angiography and Interventions, Society of Cardiovascular Anesthesiologists, and Society of Vascular Medicine Endorsed by the Society of Hospital Medicine. J Nucl Cardiol. 2015 Feb;22(1):162-215. doi: 10.1007/s12350-014-0025-z. No abstract available. PMID 25523415
- [Background] Hawn MT, Graham LA, Richman JS, Itani KM, Henderson WG, Maddox TM. Risk of major adverse cardiac events following noncardiac surgery in patients with coronary stents. JAMA. 2013 Oct 9;310(14):1462-72. doi: 10.1001/jama.2013.278787. PMID 24101118
- [Background] Brilakis ES, Banerjee S. Patient with coronary stents needs surgery: what to do? JAMA. 2013 Oct 9;310(14):1451-2. doi: 10.1001/jama.2013.279123. No abstract available. PMID 24101010
- [Background] Luckie M, Khattar RS, Fraser D. Non-cardiac surgery and antiplatelet therapy following coronary artery stenting. Heart. 2009 Aug;95(16):1303-8. doi: 10.1136/hrt.2008.161273. Epub 2009 Feb 12. PMID 19218260
- [Background] Palmerini T, Biondi-Zoccai G, Della Riva D, Mariani A, Genereux P, Branzi A, Stone GW. Stent thrombosis with drug-eluting stents: is the paradigm shifting? J Am Coll Cardiol. 2013 Nov 19;62(21):1915-1921. doi: 10.1016/j.jacc.2013.08.725. Epub 2013 Sep 11. PMID 24036025
- [Background] Mehran R, Rao SV, Bhatt DL, Gibson CM, Caixeta A, Eikelboom J, Kaul S, Wiviott SD, Menon V, Nikolsky E, Serebruany V, Valgimigli M, Vranckx P, Taggart D, Sabik JF, Cutlip DE, Krucoff MW, Ohman EM, Steg PG, White H. Standardized bleeding definitions for cardiovascular clinical trials: a consensus report from the Bleeding Academic Research Consortium. Circulation. 2011 Jun 14;123(23):2736-47. doi: 10.1161/CIRCULATIONAHA.110.009449. No abstract available. PMID 21670242
- [Background] Mehran R, Baber U, Steg PG, Ariti C, Weisz G, Witzenbichler B, Henry TD, Kini AS, Stuckey T, Cohen DJ, Berger PB, Iakovou I, Dangas G, Waksman R, Antoniucci D, Sartori S, Krucoff MW, Hermiller JB, Shawl F, Gibson CM, Chieffo A, Alu M, Moliterno DJ, Colombo A, Pocock S. Cessation of dual antiplatelet treatment and cardiac events after percutaneous coronary intervention (PARIS): 2 year results from a prospective observational study. Lancet. 2013 Nov 23;382(9906):1714-22. doi: 10.1016/S0140-6736(13)61720-1. Epub 2013 Sep 1. PMID 24004642
- [Background] Singla S, Sachdeva R, Uretsky BF. The risk of adverse cardiac and bleeding events following noncardiac surgery relative to antiplatelet therapy in patients with prior percutaneous coronary intervention. J Am Coll Cardiol. 2012 Nov 13;60(20):2005-16. doi: 10.1016/j.jacc.2012.04.062. Epub 2012 Oct 17. PMID 23083781
- [Background] Chalhoub V, Pottecher J, Asehnoune K, Mazoit JX, Duranteau J, Benhamou D. Cytokine response and reactive oxygen species production after low- and intermediate-risk surgery. Acta Anaesthesiol Scand. 2011 May;55(5):549-57. doi: 10.1111/j.1399-6576.2011.02419.x. Epub 2011 Mar 21. PMID 21418155
- [Background] Brilakis ES, Banerjee S, Berger PB. Perioperative management of patients with coronary stents. J Am Coll Cardiol. 2007 Jun 5;49(22):2145-50. doi: 10.1016/j.jacc.2007.02.046. Epub 2007 May 23. PMID 17543633
- [Background] Saia F, Belotti LM, Guastaroba P, Berardini A, Rossini R, Musumeci G, Tarantini G, Campo G, Guiducci V, Tarantino F, Menozzi A, Varani E, Santarelli A, Tondi S, De Palma R, Rapezzi C, Marzocchi A. Risk of Adverse Cardiac and Bleeding Events Following Cardiac and Noncardiac Surgery in Patients With Coronary Stent: How Important Is the Interplay Between Stent Type and Time From Stenting to Surgery? Circ Cardiovasc Qual Outcomes. 2016 Jan;9(1):39-47. doi: 10.1161/CIRCOUTCOMES.115.002155. Epub 2015 Dec 8. PMID 26646819
- [Background] Capodanno D, Musumeci G, Lettieri C, Limbruno U, Senni M, Guagliumi G, Valsecchi O, Angiolillo DJ, Rossini R. Impact of bridging with perioperative low-molecular-weight heparin on cardiac and bleeding outcomes of stented patients undergoing non-cardiac surgery. Thromb Haemost. 2015 Aug;114(2):423-31. doi: 10.1160/TH14-12-1057. Epub 2015 May 28. PMID 26017898
- [Background] Brilakis ES, Banerjee S. Perioperative management of drug-eluting stents: the Achilles heel of bridging. Catheter Cardiovasc Interv. 2013 Dec 1;82(7):1113-4. doi: 10.1002/ccd.25243. No abstract available. PMID 24255030
- [Background] Rossini R, Capodanno D, Lettieri C, Musumeci G, Nijaradze T, Romano M, Lortkipanidze N, Cicorella N, Biondi Zoccai G, Sirbu V, Izzo A, Guagliumi G, Valsecchi O, Gavazzi A, Angiolillo DJ. Prevalence, predictors, and long-term prognosis of premature discontinuation of oral antiplatelet therapy after drug eluting stent implantation. Am J Cardiol. 2011 Jan 15;107(2):186-94. doi: 10.1016/j.amjcard.2010.08.067. PMID 21211596
- [Background] Gerber Y, Rihal CS, Sundt TM 3rd, Killian JM, Weston SA, Therneau TM, Roger VL. Coronary revascularization in the community. A population-based study, 1990 to 2004. J Am Coll Cardiol. 2007 Sep 25;50(13):1223-9. doi: 10.1016/j.jacc.2007.06.022. Epub 2007 Sep 10. PMID 17888838
- [Background] Go AS, Mozaffarian D, Roger VL, Benjamin EJ, Berry JD, Blaha MJ, Dai S, Ford ES, Fox CS, Franco S, Fullerton HJ, Gillespie C, Hailpern SM, Heit JA, Howard VJ, Huffman MD, Judd SE, Kissela BM, Kittner SJ, Lackland DT, Lichtman JH, Lisabeth LD, Mackey RH, Magid DJ, Marcus GM, Marelli A, Matchar DB, McGuire DK, Mohler ER 3rd, Moy CS, Mussolino ME, Neumar RW, Nichol G, Pandey DK, Paynter NP, Reeves MJ, Sorlie PD, Stein J, Towfighi A, Turan TN, Virani SS, Wong ND, Woo D, Turner MB; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Executive summary: heart disease and stroke statistics--2014 update: a report from the American Heart Association. Circulation. 2014 Jan 21;129(3):399-410. doi: 10.1161/01.cir.0000442015.53336.12. No abstract available. PMID 24446411
- [Background] Rossini R, Musumeci G, Visconti LO, Bramucci E, Castiglioni B, De Servi S, Lettieri C, Lettino M, Piccaluga E, Savonitto S, Trabattoni D, Capodanno D, Buffoli F, Parolari A, Dionigi G, Boni L, Biglioli F, Valdatta L, Droghetti A, Bozzani A, Setacci C, Ravelli P, Crescini C, Staurenghi G, Scarone P, Francetti L, D'Angelo F, Gadda F, Comel A, Salvi L, Lorini L, Antonelli M, Bovenzi F, Cremonesi A, Angiolillo DJ, Guagliumi G; Italian Society of Invasive Cardiology (SICI-GISE); Italian Association of Hospital Cardiologists (ANMCO); Italian Society for Cardiac Surgery (SICCH); Italian Society of Vascular and Endovascular Surgery (SICVE); Italian Association of Hospital Surgeons (ACOI); Italian Society of Surgery (SIC); Italian Society of Anaesthesia and Intensive Care Medicine (SIAARTI); Lombard Society of Surgery (SLC); Italian Society of Maxillofacial Surgery (SICMF); Italian Society of Reconstructive Plastic Surgery and Aesthetics (SICPRE); Italian Society of Thoracic Surgeons (SICT); Italian Society of Urology (SIU); Italian Society of Orthopaedics and Traumatology (SIOT); Italian Society of Periodontology (SIdP); Italian Federation of Scientific Societies of Digestive System Diseases Lombardia (FISMAD); Association of Obstetricians Gynaecologists Italian Hospital Lombardia (AOGOI); Society of Ophthalmology Lombardia (SOL). Perioperative management of antiplatelet therapy in patients with coronary stents undergoing cardiac and non-cardiac surgery: a consensus document from Italian cardiological, surgical and anaesthesiological societies. EuroIntervention. 2014 May;10(1):38-46. doi: 10.4244/EIJV10I1A8. PMID 24832636
- [Background] Savonitto S, D'Urbano M, Caracciolo M, Barlocco F, Mariani G, Nichelatti M, Klugmann S, De Servi S. Urgent surgery in patients with a recently implanted coronary drug-eluting stent: a phase II study of 'bridging' antiplatelet therapy with tirofiban during temporary withdrawal of clopidogrel. Br J Anaesth. 2010 Mar;104(3):285-91. doi: 10.1093/bja/aep373. Epub 2010 Jan 3. PMID 20047898
- [Background] Rassi AN, Blackstone E, Militello MA, Theodos G, Cavender MA, Sun Z, Ellis SG, Cho L. Safety of "bridging" with eptifibatide for patients with coronary stents before cardiac and non-cardiac surgery. Am J Cardiol. 2012 Aug 15;110(4):485-90. doi: 10.1016/j.amjcard.2012.04.016. Epub 2012 May 15. PMID 22591672
- [Background] Warshauer J, Patel VG, Christopoulos G, Kotsia AP, Banerjee S, Brilakis ES. Outcomes of preoperative bridging therapy for patients undergoing surgery after coronary stent implantation: a weighted meta-analysis of 280 patients from eight studies. Catheter Cardiovasc Interv. 2015 Jan 1;85(1):25-31. doi: 10.1002/ccd.25507. Epub 2014 May 6. PMID 24740634
- [Background] Barra ME, Fanikos J, Gerhard-Herman MD, Bhatt DL. Bridging Experience With Eptifibatide After Stent Implantation. Crit Pathw Cardiol. 2016 Sep;15(3):82-8. doi: 10.1097/HPC.0000000000000084. PMID 27465001
- [Background] Waldron NH, Dallas T, Erhunmwunsee L, Wang TY, Berry MF, Welsby IJ. Bleeding risk associated with eptifibatide (Integrilin) bridging in thoracic surgery patients. J Thromb Thrombolysis. 2017 Feb;43(2):194-202. doi: 10.1007/s11239-016-1441-5. PMID 27798792
- [Background] Walker EA, Dager WE. Bridging with Tirofiban during Oral Antiplatelet Interruption: A Single-Center Case Series Analysis Including Patients on Hemodialysis. Pharmacotherapy. 2017 Aug;37(8):888-892. doi: 10.1002/phar.1956. Epub 2017 Jul 6. PMID 28543216
- [Background] Stern G, Rimsans J, Qamar A, Vaduganathan M, Bhatt DL. Contemporary parenteral antiplatelet bridging strategies: a single-centre real-world experience at a tertiary care centre. EuroIntervention. 2018 Jun 8;14(3):e333-e335. doi: 10.4244/EIJ-D-18-00036. No abstract available. PMID 29537373
- [Background] Urban P, Meredith IT, Abizaid A, Pocock SJ, Carrie D, Naber C, Lipiecki J, Richardt G, Iniguez A, Brunel P, Valdes-Chavarri M, Garot P, Talwar S, Berland J, Abdellaoui M, Eberli F, Oldroyd K, Zambahari R, Gregson J, Greene S, Stoll HP, Morice MC; LEADERS FREE Investigators. Polymer-free Drug-Coated Coronary Stents in Patients at High Bleeding Risk. N Engl J Med. 2015 Nov 19;373(21):2038-47. doi: 10.1056/NEJMoa1503943. Epub 2015 Oct 14. PMID 26466021
- [Background] Budaj A. Bleeding and Quality of Life. J Am Coll Cardiol. 2016 Jan 5;67(1):66-8. doi: 10.1016/j.jacc.2015.10.035. No abstract available. PMID 26764068
- [Background] Weinstein MC, Stason WB. Foundations of cost-effectiveness analysis for health and medical practices. N Engl J Med. 1977 Mar 31;296(13):716-21. doi: 10.1056/NEJM197703312961304. PMID 402576
- [Background] Cutlip DE, Windecker S, Mehran R, Boam A, Cohen DJ, van Es GA, Steg PG, Morel MA, Mauri L, Vranckx P, McFadden E, Lansky A, Hamon M, Krucoff MW, Serruys PW; Academic Research Consortium. Clinical end points in coronary stent trials: a case for standardized definitions. Circulation. 2007 May 1;115(17):2344-51. doi: 10.1161/CIRCULATIONAHA.106.685313. PMID 17470709
- [Background] Nalysnyk L, Fahrbach K, Reynolds MW, Zhao SZ, Ross S. Adverse events in coronary artery bypass graft (CABG) trials: a systematic review and analysis. Heart. 2003 Jul;89(7):767-72. doi: 10.1136/heart.89.7.767. PMID 12807853
- [Background] Angiolillo DJ, Firstenberg MS, Price MJ, Tummala PE, Hutyra M, Welsby IJ, Voeltz MD, Chandna H, Ramaiah C, Brtko M, Cannon L, Dyke C, Liu T, Montalescot G, Manoukian SV, Prats J, Topol EJ; BRIDGE Investigators. Bridging antiplatelet therapy with cangrelor in patients undergoing cardiac surgery: a randomized controlled trial. JAMA. 2012 Jan 18;307(3):265-74. doi: 10.1001/jama.2011.2002. PMID 22253393